CLINICAL TRIAL: NCT04380519
Title: An International, Multicenter, Randomized, Double-blind, Adaptive Placebo-controlled Study of the Efficacy and Safety of a Single Administration of Olokizumab and RPH-104 With Standard Therapy in Patients With Severe SARS-CoV-2 Infection (COVID-19)
Brief Title: Study of the Efficacy and Safety of a Single Administration of Olokizumab and RPH-104 With Standard Therapy in Patients With Severe Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Infection (COVID-19)
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: R-Pharm International, LLC (Industry)
Collaborators: Data Management 365 (Industry); K-Research, LLC (Industry)
Responsible Party: Sponsor
Organization: R-Pharm (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CL04041078
Record Dates: First submitted 2020-05-06; First posted 2020-05-08 (Actual); Results first posted 2022-01-24 (Actual); Last update posted 2022-01-24 (Actual); Status verified 2022-01

CONDITIONS: COVID-19
Keywords: SARS-CoV-2; Severe acute respiratory syndrome coronavirus 2; 2019-nCoV; 2019 novel coronavirus; Respiratory disease; lung disease; COVID-19; coronavirus
MeSH Terms: conditions — COVID-19; Respiration Disorders; Lung Diseases; Coronavirus Infections | interventions — olokizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- RPH -104 80 mg (Experimental): Subject randomized to receive subcutaneous single injection of 2 ml solution of RPH-104 on Day 1, in addition to standard therapy
  Interventions: Drug: RPH-104 80 mg
- Olokizumab 64 mg (Experimental): Subject randomized to receive subcutaneous single injection of 0,4 ml solution of Olokizumab on Day 1, in addition to standard therapy
  Interventions: Drug: Olokizumab 64 mg
- Placebo (Placebo Comparator): Subject randomized to receive subcutaneous single injection of 2 ml solution of Placebo on Day 1, in addition to standard therapy
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RPH-104 80 mg — solution for subcutaneous administration 40 mg/mL, 2 mL in the 4-mL glass vial
  Arms: RPH -104 80 mg
Drug: Olokizumab 64 mg — solution for subcutaneous administration 160 mg/mL, in the 2-mL glass vial (target volume 0,4 ml)
  Arms: Olokizumab 64 mg
Drug: Placebo — Normal Saline (0.9% Sodium Chloride solution for Injection), in the market package
  Arms: Placebo

SUMMARY:
The primary objective of the study was to evaluate the efficacy and safety of a single dose of RPH-104 (80 mg) or OKZ (64 mg) compared to placebo in addition to standard therapy in patients with severe SARS-CoV-2 infection (COVID-19) at Day 15 of the study.

DETAILED DESCRIPTION:
The study consisted of two phases:

* Pilot phase: the first 189 patients were randomized in three groups to receive OKZ, RPH-104 (63 patients per group), followed by an interim analysis of efficacy and safety data.
* The main phase was the conduct of all procedures prespecified in the protocol. Based on results of interim analysis no changes were made regarding the sample size or primary efficacy endpoint.

For each patient the study included the following periods:

* Screening period for no more than 48 hours before the start of the day of randomization (Day 1). During the screening period, an assessment was performed to determine whether the patient met the eligibility criteria;
* Treatment period lasting from the end of the screening (considered as the beginning of the Day 1) to 23:59 of the Day 1, including randomization of the patients in the treatment groups and then a single administration of the study drug;
* Follow-up period lasting from 00:00 of the Day 2 to 23:59 of the Day 29, including an assessment of the efficacy and safety after administration of the study drug.

Eligible patients were randomized to one of three treatment groups to receive a single subcutaneous injection: RPH-104 80 mg, OKZ 64 mg or placebo in addition to standard care for patients with COVID-19 as per the routine practice in participating facilities. Further, during the term of hospitalization, the clinical observation was performed (Day 1 - Day 15 of the Last Hospitalization Day (LHD), whichever comes first). This was followed by a follow-up period from the from Day 15 or LHD (whichever comes first) to Day 29.

Standard COVID-19 therapy, as per the institution routine practice, was permitted during the study, except the prohibited protocol medication (during the whole period of the study) and tocilizumab and sarilumab (during the first 24 hours after the study treatment administration).

In the absence of positive dynamics in the patient's condition (as per Investigator's judgement), it was possible to administrate a single dose of tocilizumab or sarilumab (in accordance with the actual recommendations), after the 24 hours from one of the study drug's administration.

On Day 15 primary endpoint of patient's clinical status (response to the study therapy) was assessed. The response to the therapy was considered as improvement of the patient's clinical status by at least 1 point on a 6-point COVID-19 scale in the absence of tocilizumab or sarilumab administration.

The last patient's visit in the study was the visit on Day 29. If the patient was discharged from the hospital earlier than Day 15 or Day 29, patient's clinical status at these visits were assessed by phone call.

The total expected duration of the study for each patient was not more than 31 days, including 48 hours of screening, 1 day of the study drug administration and 28 days of observation.

ELIGIBILITY:
Inclusion criteria:

1. The presence of a voluntarily signed and dated Patient Informed Consent Form for participation in this study, or a record of an Medical Consilium decision justifying patient's participation in case of patient is unable to state his/her will.
2. Having either of the following COVID-associated respiratory syndromes:

   * pneumonia with oxygenation saturation SpO2 ≤93% (on room air) or respiratory rate greater than 30/min;
   * Acute respiratory distress syndrome (ARDS) ( PaO2/FiO2 ≤ 300 mmHg or SpO2/FiO2 ≤ 315 if PaO2 is not available).
3. COVID-19 diagnosis based on:

   * laboratory-confirmed SARS-CoV-2 infection as determined by Polymerase Chain Reaction method (PCR).

OR

• Bilateral changes in the lungs typical for COVID-19, based on chest computed tomography results.

Exclusion criteria:

1. A history of hypersensitivity to the study drugs (RPH-104 and/or OKZ), and/or their components.
2. The presence of any of the following laboratory abnormalities:

   * absolute neutrophil counts < 0.5 x 10^9 L
   * white blood cell count < 2 x 10^9 L
   * platelet count <50 x 10^9 L
   * Alanine aminotransferase (ALT) and/or Aspartate aminotransferase (AST) ≥ 3.0 x Upper Limit of Normal (ULN)
3. Severe renal failure: creatinine clearance < 30 mL/min
4. Septic shock (vasopressors are required to maintain mean arterial pressure ≥ 65 mm Hg and lactate ≥ 2 mmol/L in the absence of hypovolemia)
5. The disease progresses to death over the next 24 hours, regardless of treatment, according to Investigator.
6. Perforation of the gastrointestinal tract, a history of diverticulitis.
7. Administration of plasma from COVID-19 convalescent donors within 4 weeks before study enrollment and/or planned administration during the study.
8. Recent (less then 5 half-lives) administration of tocilizumab or sarilumab;
9. Recent (less then 5 half-lives) or planned during the current study period use of the following drugs:

   * biologics (except RPH-104 or OKZ) with immunosuppressive effect, including, but not limited to: Interleukin-1 (IL-1) inhibitors (anakinra, rilonacept, canakinumab), IL- 6 inhibitors (except tocilizumab and sarilumab), IL-17A inhibitors (secukinumab), tumor necrosis factor α (TNFα) inhibitors (infliximab, adalimumab, etanercept, etc.), antiB-cell drugs, etc.
   * other immunosuppressive drugs (with the exception of methotrexate in a dose of up to 25 mg/week), including, but not limited to:

     1. high doses of glucocorticoids (equivalent to prednisolone > 1 mg/kg) orally or parenterally;
     2. Janus kinase (JAK) kinase inhibitors; cyclophosphamide, etc.
10. Concurrent participation in another clinical trial.
11. Pregnancy, breastfeeding.
12. A history of active tuberculosis, or active tuberculosis suspected by the Investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Actual)
Dates: Start 2020-04-23 (Actual); Primary Completion 2020-07-10 (Actual); Study Completion 2020-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mikhail Samsonov, Study Director — Chief Medical Officer, R-Pharm
Locations (16):
- Russia (16):
  - Private healthcare institution "Clinical Hospital" Russian Railways-Medicine named after N. A. Semashko", Moscow
  - State Budget Healthcare Institution "City Clinical Hospital № 15 named after O.M. Filatov" of Moscow City Healthcare Department, Moscow
  - Federal State Budgetary Institution "Federal Center for Cerebrovascular Pathology and Stroke" of the Ministry of Health of the Russian Federation, Moscow
  - Federal State Autonomous Education Insitution of High Education the First Moscow State Medical University named after I.M. Sechenov of Ministry of Healthcare of Russian Federation (Sechenov University), Moscow
  - Federal State Autonomous Education Institution of High Education the First Moscow State Medical University named after I.M. Sechenov of Ministry of Healthcare of the Russian Federation (Sechenov University), Moscow
  - Federal State Budgetary Institution "Central Clinical Hospital with Polyclinic" of Administrative Directorate of the President of the Russian Federation, Moscow
  - Federal State Budget Institution "National Medicine Research Center on Cardiology" By Ministry of Healthcare of Russian Federation, Moscow
  - State Budget Institution of Healthcare "City Clinical Hospital #52", Moscow City Healthcare Department, Moscow
  - State budgetary healthcare institution City Clinical Hospital named after S.I. Spasokukotsky Department of Health of the city of Moscow City Clinical Hospital No. 50, Moscow
  - Moscow State Budget Institution of Healthcare "Scientific Research Institute of Emergency Medicine named after N.V. Sklifosovsky of Moscow Department of Healthcare", Moscow
  - АО "State Company "Medsi" based on Clinical Hospital №1", Moscow
  - Federal State Budgetary Educational Institution of Higher Education "Volga Research Medical University" of the Ministry of Health of the Russian Federation, Nizhny Novgorod
  - Federal Budgetary State Healthcare Institution "National Medical Research Center named after B.A. Almazov", Saint Petersburg
  - Saint-Petersburg State Budget Institution of Healthcare "City Hospital №40", Saint Petersburg
  - Budgetary Health Institution Voronezh Regional Clinical Hospital №1, Voronezh
  - State Budget Healthcare Institution of Yaroslavl Region "Yaroslavl Region Clinical Hospital of War Veterans", Yaroslavl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 16 clinical sites in Russian Federation. 381 subjects were screened and 372 subjects were enrolled (randomized). A total of 371 subjects were treated, and 336 subjects completed the study. A total of 372 subjects were analyzed for efficacy in the Intent-to-Treat (ITT) Population, 352 subjects in the modified ITT Population (mITT) and 371 subjects were analyzed for safety in the Safety Population.
Groups:
- RPH -104 80 mg: Subcutaneous single injection of RPH-104 80 mg (2 ml 40 mg/mL solution) on Day 1, in addition to standard therapy.
- Olokizumab 64 mg: Subcutaneous single injection of Olokizumab 64 mg (0,4 ml 160 mg/mL solution) on Day 1, in addition to standard therapy.
- Placebo: Subcutaneous single injection of 2 ml solution of Placebo (Normal Saline) on Day 1, in addition to standard therapy.
Period: Overall Study
Arm/Group | RPH -104 80 mg | Olokizumab 64 mg | Placebo
Started | 124 | 124 | 124
Intent-to-Treat (ITT) | 124 | 124 | 124
Modified Intent-to-Treat (mITT) | 115 | 119 | 118
Safety Population | 123 | 124 | 124
Completed | 106 | 113 | 117
Not Completed | 18 | 11 | 7
Not completed — Withdrawal by Subject | 4 | 0 | 1
Not completed — Death | 14 | 9 | 6
Not completed — Adverse Event | 0 | 1 | 0
Not completed — relatives' decision | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RPH -104 80 mg | Olokizumab 64 mg | Placebo | Total
Number analyzed (Participants) | 124 | 124 | 124 | 372
Age, Continuous [Mean (Full Range); unit: years] | 58.0 [28.0 to 92.0] | 59.6 [26.0 to 93.0] | 59.7 [29.0 to 86.0] | 59.1 [26.0 to 93.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 58 | 57 | 176
  Male | 63 | 66 | 67 | 196
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 124 | 123 | 124 | 371
  Asian | 0 | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 1
  Not Hispanic or Latino | 123 | 123 | 124 | 370
  Not reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Responders in Each Treatment Group
Description: Proportion of patients, responded to the study therapy, in each of the treatment groups.
  A responder is a patient who has not received tocilizumab or sarilumab and who has a clinical status improvement of ≥1 point on the 6-point COVID-19 scale (where 1 is the most favorable outcome and 6 is the most undesirable outcome) 15 days after the administration of the study drug:
  1. Not hospitalized, no activity limitations.
  2. Not hospitalized, limited activity.
  3. Hospitalized, not requiring supplemental oxygen.
  4. Hospitalized, supplemental oxygen with independent breathing.
  5. Hospitalized; mechanical ventilation (invasive/non-invasive) or Extracorporeal membrane oxygenation (ECMO).
  6. Death.
Time Frame: Day 15
Population: The intent-to-treat (ITT) population included all randomized patients.
Measure: Count of Participants; unit: Participants
Arm/Group | RPH -104 80 mg | Olokizumab 64 mg | Placebo
Number analyzed (Participants) | 124 | 124 | 124
Participants | 88 | 98 | 87
Statistical Analysis 1: Comparison: RPH -104 80 mg vs Placebo; Test type: Superiority; p = 0.434, Maximal Likelihood Estimator (MLE) model — Hochberg adjustment was applied for p-values; Risk Ratio (RR) = 1.012, 97.5% CI 1-sided [lower limit 0.880]
Statistical Analysis 2: Comparison: Olokizumab 64 mg vs Placebo; Test type: Superiority; p = 0.073, Maximal Likelihood Estimator (MLE) model — Hochberg adjustment was applied for p-values; Risk Ratio (RR) = 1.125, 97.5% CI 1-sided [lower limit 0.989]

2. Secondary Outcome: Change Over Time in the Clinical Status of Patients Using a 6-point Ordinal Scale
Description: Changes of patients' clinical status on a 6 points ordinal scale (where 1 was the most favorable outcome and 6 was the most undesirable outcome) over time.
  The 6-point ordinal scale included the following categories:
  1. Not hospitalized, no activity limitations.
  2. Not hospitalized, limited activity.
  3. Hospitalized, not requiring supplemental oxygen.
  4. Hospitalized, supplemental oxygen, with independent breathing.
  5. Hospitalized, mechanical ventilation (invasive/non-invasive) or ECMO.
  6. Death.
Time Frame: from Day 2 until Day 15, Day 29
Population: The ITT population was the primary analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | RPH -104 80 mg | Olokizumab 64 mg | Placebo
Number analyzed (Participants) | 124 | 124 | 124
Participants
  Day 15: improvement | 88 | 99 | 96
  Day 15: worsening (including deaths) | 13 | 8 | 7
  Day 15: without change | 15 | 11 | 17
  Day 15: no data | 8 | 6 | 4
  Day 29: improvement | 105 | 113 | 111
  Day 29: worsening (including deaths) | 14 | 9 | 8
  Day 29: without change | 1 | 0 | 1
  Day 29: no data | 4 | 2 | 4

3. Secondary Outcome: The Proportion of Patients With an Improvement in Clinical Status by 2 or More Points on the 6-point Ordinal Scale During the Study With no Use of Tocilizumab or Sarilumab
Description: The proportion of patients with an improvement in clinical status by 2 or more points on the 6-point ordinal scale (where 1 was the most favorable outcome and 6 was the most undesirable outcome) during the study with no use of tocilizumab or sarilumab.
  The 6-point ordinal scale included the following categories:
  1. Not hospitalized, no activity limitations.
  2. Not hospitalized, limited activity.
  3. Hospitalized, not requiring supplemental oxygen.
  4. Hospitalized, supplemental oxygen, with independent breathing.
  5. Hospitalized, mechanical ventilation (invasive/non-invasive) or ECMO.
  6. Death.
Time Frame: Day 29
Population: The ITT population was the primary analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | RPH -104 80 mg | Olokizumab 64 mg | Placebo
Number analyzed (Participants) | 124 | 124 | 124
Participants | 94 | 103 | 94
Statistical Analysis 1: Comparison: RPH -104 80 mg vs Placebo; Test type: Superiority; p = 0.393, Maximal Likelihood Estimator (MLE) model — unadjusted; Risk Ratio (RR) = 1.019, 97.5% CI 1-sided [lower limit 0.892]
Statistical Analysis 2: Comparison: Olokizumab 64 mg vs Placebo; Test type: Superiority; p = 0.061, Maximal Likelihood Estimator (MLE) model — unadjusted; Risk Ratio (RR) = 1.098, 97.5% CI 1-sided [lower limit 0.975]

4. Secondary Outcome: The Proportion of Patients Who Received Tocilizumab or Sarilumab for COVID-19 During the Study
Description: The proportion of patients who received tocilizumab or sarilumab for COVID-19 during the study
Time Frame: from Day 2 until the Day 29
Population: The ITT population was the primary analysis population.
Measure: Count of Participants; unit: Participants
Arm/Group | RPH -104 80 mg | Olokizumab 64 mg | Placebo
Number analyzed (Participants) | 124 | 124 | 124
Participants | 10 | 5 | 15
Statistical Analysis 1: Comparison: RPH -104 80 mg vs Placebo; Test type: Superiority; Risk Ratio (RR) = 0.67, 95% CI 2-sided [0.31 to 1.44]
Statistical Analysis 2: Comparison: Olokizumab 64 mg vs Placebo; Test type: Superiority; Risk Ratio (RR) = 0.33, 95% CI 2-sided [0.12 to 0.89]
Statistical Analysis 3: Comparison: RPH -104 80 mg vs Placebo; Test type: Superiority; Odds Ratio (OR) = 0.64, 95% CI 2-sided [0.28 to 1.49]
Statistical Analysis 4: Comparison: Olokizumab 64 mg vs Placebo; Test type: Superiority; Odds Ratio (OR) = 0.31, 95% CI 2-sided [0.11 to 0.87]

5. Secondary Outcome: Mortality Rate During the Study
Description: Mortality rate over the follow-up period of the study
Time Frame: from Day 1 until Day 29
Population: The safety population included all patients who received the IP (371 patients: 124 patients in the OKZ group, 123/124 (99.2%) patients in the RPH-104 group (1 patient did not received the IP) and 124 patients in the Placebo group).
Measure: Count of Participants; unit: Participants
Arm/Group | RPH -104 80 mg | Olokizumab 64 mg | Placebo
Number analyzed (Participants) | 123 | 124 | 124
Participants | 14 | 9 | 6
Statistical Analysis 1: Comparison: RPH -104 80 mg vs Placebo; Test type: Superiority; Risk Ratio (RR) = 2.35, 95% CI 2-sided [0.93 to 5.92]
Statistical Analysis 2: Comparison: Olokizumab 64 mg vs Placebo; Test type: Superiority; Risk Ratio (RR) = 1.5, 95% CI 2-sided [0.55 to 4.09]
Statistical Analysis 3: Comparison: RPH -104 80 mg vs Placebo; Test type: Superiority; Odds Ratio (OR) = 2.53, 95% CI 2-sided [0.94 to 6.81]
Statistical Analysis 4: Comparison: Olokizumab 64 mg vs Placebo; Test type: Superiority; Odds Ratio (OR) = 1.54, 95% CI 2-sided [0.53 to 4.46]

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs), except serious ones, were recorded from the moment of the use of the IP. AEs recorded prior to the start of the study therapy, but after the patient was included in the study, were recorded in the electronic CRF Case report form (eCRF) as "Concomitant diseases". AEs were registered until the end of the follow-up period (day 29).
Description: All AE analyses were performed in the safety population. (The safety population included all patients who received the IP.) No statistical comparisons were conducted on the AE data. Data for treatment-emergent AEs (TEAEs) were reported below. TEAE is an AE that started at or after the time of administration of the randomized IP.
Arm/Group | RPH -104 80 mg | Olokizumab 64 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 14/123 | 9/124 | 6/124
Serious Adverse Events (participants affected / at risk) | 15/123 | 10/124 | 8/124
Other Adverse Events (participants affected / at risk) | 30/123 | 23/124 | 35/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RPH -104 80 mg (N=123) | Olokizumab 64 mg (N=124) | Placebo (N=124)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Sepsis (Infections and infestations) | 3 (3) | 2 (2) | 3 (3)
Septic shock (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Viral sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1)
Pneumothorax spontaneous (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RPH -104 80 mg (N=123) | Olokizumab 64 mg (N=124) | Placebo (N=124)
Alanine aminotransferase increased (Investigations) | 13 (13) | 11 (11) | 15 (15)
Aspartate aminotransferase increased (Investigations) | 12 (12) | 9 (9) | 12 (12)
Gamma-glutamyltransferase increased (Investigations) | 5 (5) | 3 (3) | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any study related information could be made public available only after Sponsors written permission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-04-26): https://cdn.clinicaltrials.gov/large-docs/19/NCT04380519/Prot_SAP_000.pdf